CLINICAL TRIAL: NCT05498610
Title: Investigation of Pharmacokinetic Properties of Subcutaneously co Administered Single Doses of NNC0480-0389 and Semaglutide in Healthy Chinese Male Subjects
Brief Title: A Research Study of How the Medicine NNC0480-0389 Taken With Semaglutide Works in the Body of Healthy Chinese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9389-4774; U1111-1264-4516 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1.7 mg NNC0408-0389 plus 0.5 mg semaglutide (Experimental): Participants will receive a single subcutanous dose of 1.7 mg of NNC0408-0389 in combination with a fixed dose of 0.5 mg semaglutide administered as separate injections
  Interventions: Drug: NNC0480 0389; Drug: Semaglutide
- 8.6 mg NNC0480-0389 plus 0.5 mg semaglutide (Experimental): Participants will receive a single subcutanous dose of 8.6 mg of NNC0408-0389 in combination with a fixed dose of 0.5 mg semaglutide administered as separate injections
  Interventions: Drug: NNC0480 0389; Drug: Semaglutide
- 30 mg NNC0480 0389 plus 0.5 mg semaglutide (Experimental): Participants will receive a single subcutanous dose of 30 mg of NNC0408-0389 in combination with a fixed dose of 0.5 mg semaglutide administered as separate injections
  Interventions: Drug: NNC0480 0389; Drug: Semaglutide

INTERVENTIONS:
Drug: NNC0480 0389 — Participants will get 1 injections of NNC04800389. It will be injected with a needle into a skin fold on the abdomen.
  The study will last for a maximum of 72 days
Drug: Semaglutide — Participants will get 1 injections of semaglutide. It will be injected with a needle into a skin fold on the abdomen.
  The study will last for a maximum of 72 days

SUMMARY:
This study looks at how the new medicine called NNC0480-0389 works in the body of Chinese men when it is given at different doses together with a fixed dose of semaglutide. Participants will get one injection of NNC0480-0389 and one injection of semaglutide - which dose of NNC0480-0389 participants get is decided by chance.

NNC0480-0389 is a new medicine that has not been previously approved. It means that the medicine has not yet been approved by the health authorities.

Semaglutide is a newly approved antidiabetic medicine that helps to lower blood sugar levels in people with type 2 diabetes.

NNC0480-0389 is being developed to be given together with semaglutide. NNC0480-0389 targets a different part of the system that regulates sugar levels in the body than semaglutide. Therefore, it is expected that together NNC0480-0389 and semaglutide will more effectively lower sugar levels in the blood in people with type 2 diabetes.

Participants will get 2 injections of the study medicine (one of each). It will be injected with a needle into a skin fold on participants abdomen.

The study will last for a maximum of 72 days. Partcicipants will have 10 scheduled visits with the study doctor. For 1 of the visits participants will stay at the clinic for 6 days (5 nights). The study includes blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male participants aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 20.0 kg/m^2 and 27.9 kg/m^2 (both inclusive).
* Body weight equal to or greather than 54.0 kg.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Any disorder which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Glycated haemoglobin (HbA1c) geather han or equal to 6.5 % (48 mmol/mol) at screening.
* Use of prescription medicinal products or non-prescription drugs (including Chinese traditional medicine or local medicine), except routine vitamins, occasional use of paracetamol, ibuprofen and acetylsalicylic acid, or topical medication not reaching systemic circulation, within 14 days before screening.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
AUC0-∞,NNC0480-0389,SD Area under the NNC0480-0389 plasma concentration-time curve from time 0 to infinity after a single dose (SD) | From pre-dose (day 1) to completion of the post-dose follow-up visit (day 43)
  measured in hnmol^L
Cmax,NNC0480-0389,SD Maximum plasma concentration of NNC0480-0389 after a single dose | From pre-dose (day 1) to completion of the post-dose follow-up visit (day 43)
  measured in nmol/L

SECONDARY OUTCOMES:
AUC0-∞,sema,SD Area under the semaglutide plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (day 1) to completion of the post-dose follow-up visit (day 43)
  measured in hnmol^L
Cmax,sema,SD The maximum plasma concentration of semaglutide after a single dose | From pre-dose (day 1) to completion of the post-dose follow-up visit (day 43)
  measured in nmol^L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com